CLINICAL TRIAL: NCT04987710
Title: Intracranial Rescue Stenting for Acute Ischemic Stroke, Predictors of Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mohammed Hamdy Ghazally, Assistant lecturer, Assiut University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRSFAIS-POO
Record Dates: First submitted 2021-07-17; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Ischemic Stroke; Thromboembolic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: intracranial rescue stenting — use of intracranial rescue stenting as re-perfusion technique after failed thrombectomy

SUMMARY:
The use of rescue intracranial stenting is thought to be associated with better outcomes than with patients received medical treatment only after failed thrombectomy as Reperfusion technique. This raised the questions about the factors that affect outcomes of rescue intracranial stenting angioplasty, so the best outcomes can be achieved.

DETAILED DESCRIPTION:
Mechanical Thrombectomy is the first line therapy in acute ischemic stroke due to large vessel occlusion. Recently, there is an increasing number of patients with failed re perfusion after mechanical thrombectomy, due to preexisting high degree of intracranial stenosis or failed mechanical thrombectomy. This is associated with poor clinical and functional outcome for the patients.

The percentage of patients with failed mechanical thrombectomy is as high as 40-45% of all patients with ischemic stroke due to large vessel occlusion.

This group is in need for rescue intracranial stenting to achieve re-canalization of the occluded vessel and restore perfusion.

The results demonstrated superiority of medical management over stenting with less complications and this had almost put the intracranial stenting to rest for years.

The main complication related to rescue stenting are ischemic complications especially thromboembolic events related to thrombus detachment, symptomatic intracerebral hemorrhage and re-stenosis of cerebral arteries after stenting.

Recently, the results of the Chinese Angioplasty and Stenting for Symptomatic Intracranial Severe Stenosis trial and the Wingspan Stent System Post Market Surveillance Study (WEAVE trial) showed that most of complications are related to peri-procedural techniques. This raise the interest again in the efficacy of intracranial stenting as treatment modality for selected patients.

The use of rescue intracranial stenting is thought to be associated with better outcomes than with patients received medical treatment only after failed thrombectomy as Reperfusion technique. This raised the questions about the factors that affect outcomes of rescue intracranial stenting angioplasty, so the best outcomes can be achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute ischemic stroke due to large vessel occlusion as confirmed by CT angiography or Magnetic resonance (MR) angiography.
2. Baseline NIHSS >6.
3. Presenting within the first 6 hours from onset of symptoms.
4. First ever stroke or pre-stroke modified Rankin Score (mRS) ≤1.

Exclusion Criteria:

1. Patients with intra cranial hemorrhage.
2. Patients younger than 18 years.
3. Patients with acute ischemic stroke due to small vessel disease or vasculitis.
4. Patients with acute ischemic stroke due to occlusion of vessels of posterior circulation.
5. Patients who refused to be included in the study.
6. Patients with contraindications to intracranial stent placement (as total occlusion of artery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
number of participants with good re-perfusion after successful rescue stenting | 12 months
  this may help in case selection for best outcomes of the procedure

SECONDARY OUTCOMES:
Compare the clinical outcomes of participants with rescue stenting with those who received medical treatment. | 12 months
Compare the radio-logical outcomes of participants with rescue stenting with those who received medical treatment. | 12 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campbell BC, Mitchell PJ; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2365-6. doi: 10.1056/NEJMc1504715. No abstract available. PMID 26061843
- [Background] Behme D, Weber W, Mpotsaris A. Acute Basilar Artery Occlusion with Underlying High-Grade Basilar Artery Stenosis: Multimodal Endovascular Therapy in a Series of Seven Patients. Clin Neuroradiol. 2015 Sep;25(3):267-74. doi: 10.1007/s00062-014-0303-9. Epub 2014 Apr 12. PMID 24727890
- [Background] Gao F, Lo WT, Sun X, Mo DP, Ma N, Miao ZR. Combined Use of Mechanical Thrombectomy with Angioplasty and Stenting for Acute Basilar Occlusions with Underlying Severe Intracranial Vertebrobasilar Stenosis: Preliminary Experience from a Single Chinese Center. AJNR Am J Neuroradiol. 2015 Oct;36(10):1947-52. doi: 10.3174/ajnr.A4364. Epub 2015 Jun 18. PMID 26089317
- [Background] Stracke CP, Fiehler J, Meyer L, Thomalla G, Krause LU, Lowens S, Rothaupt J, Kim BM, Heo JH, Yeo LLL, Andersson T, Kabbasch C, Dorn F, Chapot R, Hanning U. Emergency Intracranial Stenting in Acute Stroke: Predictors for Poor Outcome and for Complications. J Am Heart Assoc. 2020 Mar 3;9(5):e012795. doi: 10.1161/JAHA.119.012795. Epub 2020 Mar 3. PMID 32122218
- [Background] Kim GE, Yoon W, Kim SK, Kim BC, Heo TW, Baek BH, Lee YY, Yim NY. Incidence and Clinical Significance of Acute Reocclusion after Emergent Angioplasty or Stenting for Underlying Intracranial Stenosis in Patients with Acute Stroke. AJNR Am J Neuroradiol. 2016 Sep;37(9):1690-5. doi: 10.3174/ajnr.A4770. Epub 2016 Apr 14. PMID 27079369
- [Background] Baracchini C, Farina F, Soso M, Viaro F, Favaretto S, Palmieri A, Kulyk C, Ballotta E, Nico L, Cester G, Causin F. Stentriever Thrombectomy Failure: A Challenge in Stroke Management. World Neurosurg. 2017 Jul;103:57-64. doi: 10.1016/j.wneu.2017.03.070. Epub 2017 Mar 24. PMID 28347898
- [Background] Gruber P, Garcia-Esperon C, Berberat J, Kahles T, Hlavica M, Anon J, Diepers M, Nedeltchev K, Remonda L. Neuro Elutax SV drug-eluting balloon versus Wingspan stent system in symptomatic intracranial high-grade stenosis: a single-center experience. J Neurointerv Surg. 2018 Dec;10(12):e32. doi: 10.1136/neurintsurg-2017-013699. Epub 2018 Apr 7. PMID 29627786
- [Background] Baek JH, Kim BM, Heo JH, Nam HS, Kim YD, Park H, Bang OY, Yoo J, Kim DJ, Jeon P, Baik SK, Suh SH, Lee KY, Kwak HS, Roh HG, Lee YJ, Kim SH, Ryu CW, Ihn YK, Kim B, Jeon HJ, Kim JW, Byun JS, Suh S, Park JJ, Lee WJ, Roh J, Shin BS. Number of Stent Retriever Passes Associated With Futile Recanalization in Acute Stroke. Stroke. 2018 Sep;49(9):2088-2095. doi: 10.1161/STROKEAHA.118.021320. PMID 30354993
- [Background] Yoon W, Kim SK, Park MS, Kim BC, Kang HK. Endovascular treatment and the outcomes of atherosclerotic intracranial stenosis in patients with hyperacute stroke. Neurosurgery. 2015 Jun;76(6):680-6; discussion 686. doi: 10.1227/NEU.0000000000000694. PMID 25988927
- [Background] Turan TN, Lynn MJ, Nizam A, Lane B, Egan BM, Le NA, Lopes-Virella MF, Hermayer KL, Benavente O, White CL, Brown WV, Caskey MF, Steiner MR, Vilardo N, Stufflebean A, Derdeyn CP, Fiorella D, Janis S, Chimowitz MI; SAMMPRIS Investigators. Rationale, design, and implementation of aggressive risk factor management in the Stenting and Aggressive Medical Management for Prevention of Recurrent Stroke in Intracranial Stenosis (SAMMPRIS) trial. Circ Cardiovasc Qual Outcomes. 2012 Sep 1;5(5):e51-60. doi: 10.1161/CIRCOUTCOMES.112.966911. No abstract available. PMID 22991350
- [Background] Terada T, Tsuura M, Matsumoto H, Masuo O, Yamaga H, Tsumoto T, Itakura T. Complications associated with stenting for cerebral arteries. Interv Neuroradiol. 2003 May 15;9(Suppl 1):165-9. doi: 10.1177/15910199030090S123. Epub 2004 Oct 22. PMID 20591247
- [Background] Alexander MJ, Zauner A, Chaloupka JC, Baxter B, Callison RC, Gupta R, Song SS, Yu W; WEAVE Trial Sites and Interventionalists. WEAVE Trial: Final Results in 152 On-Label Patients. Stroke. 2019 Apr;50(4):889-894. doi: 10.1161/STROKEAHA.118.023996. PMID 31125298